CLINICAL TRIAL: NCT02127112
Title: Ridge Augmentation Comparing the Clinical and Histologic Healing of a Cancellous Block Allograft Plus Optecure Containing Cortico-Cancellous Chips Versus Optecure Containing Cortico-Cancellous Chips Alone.
Brief Title: Ridge Augmentation Comparing a Block Allograft to a Demineralized Bone Matrix Allograft.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Principle Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14.0265
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Alveolar Process Defect
Keywords: Ridge Augmentation; Bone regeneration; Guided Bone Regeneration; Partially Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Block Allograft plus Matrix Allograft (Active Comparator): The positive control treatment will include a block allograft plus a demineralized bone matrix moldable allograft.
  Interventions: Procedure: Block Allograft plus Matrix Allograft; Procedure: Moldable Matrix Allograft
- Moldable Matrix Allograft (Experimental): In the test arm of the study the treatment will include a demineralized bone matrix moldable allograft.
  Interventions: Procedure: Moldable Matrix Allograft

INTERVENTIONS:
Procedure: Block Allograft plus Matrix Allograft — A cancellous block allograft plus a demineralized bone matrix allograft will be used as the positive control treatment.
  Other Names: Cancellous block allograft; Optecure + CCC
  Arms: Block Allograft plus Matrix Allograft
Procedure: Moldable Matrix Allograft — The test arm of this study will include a demineralized bone matrix allograft placed over resorbable bone pins.
  Other Names: Optecure + CCC; Resorbable bone pins

SUMMARY:
This study with compare the ridge dimension changes for a block allograft vs. a demineralized bone matrix moldable allograft.

DETAILED DESCRIPTION:
The patients' treatment will be randomly assigned by coin toss done by the mentor immediately after flap reflection. The examiner will be blinded to the treatment and will not have access to information indicating treatment assignment. The examiner will never see the patient between the time of grafting and complete healing at 4 months. The surgical procedure will consist of the reflection of a split-thickness flap to expose the alveolar ridge. Following complete exposure of the surgical site, vertical measurements will be taken with the acrylic occlusal stent in place, and horizontal measurements with a specially designed digital caliper. After initial surgical measurements, numerous cortical perforations will be performed with a round bur in the area of the augmentation. The control group will receive a block graft and bone screw for stabilization, with voids being filled by the Optecure+CCC®. The test group therapy will include graft with the Optecure+CCC® and the use of Bone Pin® for space maintenance. Horizontal dimension will be established by graft dimensions, bone screws, or bone pins when necessary, for each planned implant area. Longer span edentulous spaces will be divided into individual sites as follows: 5 mm from natural teeth to future mid-implant sites and 7 mm between two future mid-implant sites. The bone pins and bone blocks with bone screws will be placed to allow enough exposure for augmentation to achieve 9 mm horizontal width available for implant placement. Vertical and horizontal measurements will again be taken with the acrylic occlusal stent and calipers prior to flap closure. An resorbable membrane will cover both test and control groups. A monofilament suture material will be used. The surgical procedures will be documented with clinical photographs.

ELIGIBILITY:
Inclusion Criteria:

* At least a one tooth area with a ridge defect, treatment planned to receive a dental implant. The site must be bordered by at least one tooth.
* Healthy person that is at least 18 years old.
* Patient understands and signs an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

* Patients with debilitating systemic diseases, diseases that significantly affect the periodontium, or psychological problems that would interfere with treatment.
* Previous head and neck radiation or chemotherapy within the previous 12 months.
* Patients with known allergy to any of the materials that will be used in the study.
* Smokers.
* Patients who need prophylactic antibiotics prior to dental procedures.
* Patients on long-term steroid therapy or oral bisphosphonates > 3 years or any IV bisphosphonates.
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Site width (horizontal) changes by comparing the pre- to post-augmentation dimensions of hard tissues. | 4 months
  Measurement of the horizontal changes will be completed with a manual periodontal probe

SECONDARY OUTCOMES:
Site height (vertical) changes by comparing the pre- to the post-augmentation dimensions of hard tissues. | 4 months
  Measurement of of height will be used with an acrylic stent and a manual periodontal probe.
Histologic composition of the healed ridge. | 4 month
  At the time of re-entry, a trephine core specimen will be taken. This specimen will be examined under a microscope to determine the vital bone characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, MSD, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - Graduate Periodontics Clinic, University of Louisville, Louisville, Kentucky
  - U of L Dental School, Louisville, Kentucky